CLINICAL TRIAL: NCT02889900
Title: A Single Arm, Open-label, Phase IIb Study to Assess the Efficacy and Safety of the Combination of Cediranib and Olaparib Tablets in Women With Recurrent Platinum Resistant Epithelial Ovarian Cancer, Including Fallopian Tube and/or Primary Peritoneal Cancer Who do Not Carry a Deleterious or Suspected Deleterious Germline BRCA Mutation
Brief Title: Efficacy and Safety Study of Cediranib in Combination With Olaparib in Patients With Recurrent Platinum-Resistant Ovarian Cancer
Acronym: CONCERTO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Myriad Genetic Laboratories, Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8488C00001
Expanded Access: NCT03079687 (Approved for marketing)
Record Dates: First submitted 2016-07-20; First posted 2016-09-07 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Recurrent Platinum Resistant Ovarian Cancer
Keywords: ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — cediranib; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- combination of cediranib and olaparib (Experimental): Open label
  Interventions: Drug: cediranib and olaparib

INTERVENTIONS:
Drug: cediranib and olaparib — Cediranib tablets oral dose 30 mg once daily; Olaparib(Lynparza) tablet 200 mg twice daily
  Dose reduction for both products is allowed
  Other Names: Olaparib: also known as Lynparza

SUMMARY:
This is an open label, single arm, multi-center study to assess the efficacy and safety of the combination of cediranib and olaparib tablets in platinum-resistant relapsed high grade serous, high grade endometroid or clear cell ovarian, fallopian tube or primary peritoneal carcinoma patients who have received at least 3 prior lines of chemotherapy and who do not carry deleterious or suspected deleterious germline breast cancer susceptibility gene (BRCA) mutations.

DETAILED DESCRIPTION:
The study will recruit approximately 60 patients aged ≥18 years, with histologically proven diagnosis of platinum-resistant relapsed high grade serous, high grade endometroid or clear cell ovarian, fallopian tube or primary peritoneal carcinoma who have received at least 3 prior lines of therapy, and who do not carry a deleterious or suspected deleterious germline BRCA mutation. All patients should have recurrent platinum resistant disease. The receipt of prior antiangiogenic treatment (e.g. bevacizumab) is optional. If used, it can be in the first line or recurrent setting. To be eligible to enter the study, all patients should have measurable disease (as assessed by the Investigator).

There is no maximum duration for taking the study treatments (cediranib+olaparib). Patients should continue on study treatments until objective radiological disease progression, as defined by RECIST version 1.1 guidelines, or they meet other discontinuation criteria. Following discontinuation of study treatment patients will be followed for disease progression (if they have not already progressed), survival and post-progression anti cancer therapies until the data cut-off for the primary analysis, approximately 8 months after enrollment of the last patient.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to provide written informed consent, and to comply with the requirements of the protocol
2. Females aged ≥18 years with previous histologically proven diagnosis of high grade serous, high grade endometroid or clear cell ovarian cancer, fallopian tube or primary peritoneal carcinoma
3. No evidence of deleterious or suspected deleterious germline mutation in BRCA1 or BRCA2 genes
4. Recurrent platinum-resistant disease, defined as disease progression within 6 months (182 days) of the last receipt of platinum-based chemotherapy
5. CT/MRI evidence of measurable disease as per RECIST 1.1 defined as at least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) and which is suitable for accurate repeated measurements
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
7. Life expectancy ≥12 weeks
8. Prior receipt of antiangiogenic treatment, including but not limited to bevacizumab, is optional. If used, it can be used in the first line or recurrent setting.
9. At least three prior lines of therapy for advanced ovarian cancer as defined in the protocol
10. Confirmation of the availability of a tumor sample from the primary or recurrent cancer must be provided
11. Patients must have adequate organ and bone marrow function
12. Adequately controlled blood pressure
13. Adequately controlled thyroid function, with no symptoms of thyroid dysfunction
14. Able to swallow and retain oral medications and without gastrointestinal illnesses that would preclude absorption of cediranib or olaparib
15. Postmenopausal or evidence of non-childbearing status for women of childbearing potential as confirmed by a negative urine or serum pregnancy test within 7 days prior to start of IPs

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
2. Previous enrollment in the present study.
3. Exposure to any IP during the last 4 weeks prior to enrollment.
4. Previous treatment with PARP inhibitor. For this study, BSI-201 (iniparib) is not considered as PARPi
5. Recent cancer-directed therapies: Radiotherapy (RT) within 4 weeks, chemotherapy or other systemic anti-cancer therapy within 4 weeks, or prior anti-angiogenic treatment (e.g., bevacizumab) within 6 weeks prior to starting treatment
6. Cancer antigen-125 (CA-125) only disease without RECIST 1.1 measurable disease
7. Major surgical procedure within 2 weeks prior to starting treatment; patients must have recovered from any effects of any major surgery and surgical wound should have healed prior to starting treatment
8. Clinically significant signs and/or symptoms of bowel obstruction within 3 months prior to starting treatment
9. History of intra-abdominal abscess within 3 months prior to starting treatment
10. History of GI perforation. Patients with a history of abdominal fistula will be considered eligible if the fistula was surgically repaired, there has been no evidence of fistula for at least 6 months prior to starting treatment, and patient is deemed to be at low risk of recurrent fistula
11. Other malignancy within the last 5 years
12. Persisting ≥Grade 2 CTCAE toxicity (except alopecia and Grade 2 peripheral neuropathy) from previous anti-cancer treatment(s)
13. Central nervous system metastases
14. Patients with any of the following: History of myocardial infarction within 6 months prior to starting treatment; Unstable angina; Resting electrocardiogram (ECG) with clinically significant abnormal findings; New York Heart Association functional classification of III or IV
15. Left ventricular ejection fraction (LVEF) < lower limit of normal (LLN) per institutional guidelines, or <55%, if threshold for normal not otherwise specified by institutional guidelines, for patients with the following risk factors: Prior treatment with anthracyclines; Prior treatment with trastuzumab; Prior central thoracic RT, including exposure of heart to therapeutic doses of ionizing RT; History of myocardial infarction within 6-12 months prior to start of IPs; Prior history of other significant impaired cardiac function
16. History of stroke or transient ischemic attack within 6 months
17. Uncontrolled intercurrent illness
18. Patients with myelodysplastic syndrome (MDS)/ treatment-related acute myeloid leukemia (t-AML) or with features suggestive of MDS/AML
19. No prior allogenic bone marrow transplant or double umbilical cord blood transplantation
20. Known active human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C infection on antiviral treatment
21. Concomitant use of known strong or moderate CYP3A inhibitors
22. Concomitant use of known strong or moderate CYP3A inducers

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2021-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Min Lee, M.D., Principal Investigator — NIH - National Cancer Institute
Locations (24):
- United States (24):
  - Research Site, Mobile, Alabama
  - Research Site, Anchorage, Alaska
  - Research Site, Downey, California
  - Research Site, Greenbrae, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, West Hollywood, California
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Newnan, Georgia
  - Research Site, Fort Wayne, Indiana
  - Research Site, Westwood, Kansas
  - Research Site, Covington, Louisiana
  - Research Site, Towson, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Billings, Montana
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8488C00001&attachmentIdentifier=5f9ef017-7750-4f01-88a6-6dec93f6cd29&fileName=d8488c00001-csr-redacted-synopsis-errata_Redacted_2022-02-17.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with platinum-resistant relapsed high grade serous, high grade endometroid or clear cell ovarian, fallopian tube or primary peritoneal carcinoma who had received at least 3 prior lines of therapy for advanced ovarian cancer were recruited to 25 study centers in the United States in this single arm, open-label Phase IIb study.
Pre-assignment Details: Patients had no evidence of deleterious or suspected deleterious germline breast cancer susceptibility gene (gBRCA) mutations. Patients had to have measurable disease, defined as ≥1 lesion that could be assessed at baseline by computed tomography / magnetic resonance imaging and be suitable for repeated assessment.
Groups:
- Cediranib + Olaparib: Patients received a combination of cediranib 30 milligrams (mg) orally once daily (qd) and olaparib 200 mg orally twice daily (bid) until objective radiological disease progression, unacceptable toxicity or withdrawal of consent. Dose modification was allowed per protocol-defined guidelines.
Period: Overall Study
Arm/Group | Cediranib + Olaparib
Started | 62
Received Treatment | 60
Completed | 5 (Patients ongoing in study at primary analysis data cut off (DCO))
Not Completed | 57
Not completed — Adverse Event | 11
Not completed — Condition under investigation worsened | 32
Not completed — Other | 5
Not completed — Withdrawal by Subject | 7
Not completed — Not treated | 2

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) included all patients who received at least 1 dose of either of the investigational products (IPs).
Groups:
- Cediranib + Olaparib: Patients received a combination of cediranib 30 mg orally qd and olaparib 200 mg orally bid until objective radiological disease progression, unacceptable toxicity or withdrawal of consent. Dose modification was allowed per protocol-defined guidelines.
Arm/Group | Cediranib + Olaparib
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 54
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 55
  Asian | 2
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Objective Response Rate (ORR) by Independent Central Review (ICR) Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: The ORR was defined as the percentage of patients with objective response (complete response [CR] or partial response [PR]) according to RECIST 1.1 and was assessed by ICR. Only patients whose CR/PR response was confirmed by a second scan at least 4 weeks after the initial response, with no evidence of progression between the initial and CR/PR confirmation visit were included.
  CR: Disappearance of all target lesions (TLs) and non-TLs (NTLS) since baseline; any pathological lymph nodes selected as TLs must have a reduction in short axis to <10 millimeters (mm).
  PR: At least a 30% decrease in the sum of the diameters of TL, referencing the baseline sum of diameters.
  Data obtained up until progression, or last evaluable assessment in the absence of progression were included in the assessment of ORR.
Time Frame: From baseline to primary analysis DCO (8 months after last patient received their first dose of IPs). RECIST assessments were performed at baseline and every 8 weeks (+/- 1 week) after first doses of IPs until disease progression.
Population: The evaluable for response (EFR) analysis set included all patients who received at least 1 dose of IP and had measurable disease at baseline according to the independent review of baseline imaging data. RECIST assessments were performed at baseline and every 8 weeks (+/- 1 week) after first doses of IPs until disease progression.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cediranib + Olaparib
Number analyzed (Participants) | 59
percentage of patients | 15.3 [7.2 to 27.0]

2. Secondary Outcome: ORR by Investigator Assessment Using RECIST 1.1
Description: The percentage of patients with a response (CR/PR), including patients with both confirmed and unconfirmed responses, based on investigator assessed RECIST 1.1 data is presented. Confirmed responses included patients whose CR/PR response was confirmed by a second scan at least 4 weeks after the initial response, with no evidence of progression between the initial and CR/PR confirmation visit.
  CR: Disappearance of all TLs and NTLs since baseline; any pathological lymph nodes selected as TLs must have a reduction in short axis to <10 mm.
  PR: At least a 30% decrease in the sum of the diameters of TL, referencing the baseline sum of diameters.
Time Frame: as for outcome 1
Population: The FAS included all patients who received at least 1 dose of either of the IPs.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cediranib + Olaparib
Number analyzed (Participants) | 60
percentage of patients | 26.7 [16.1 to 39.7]

3. Secondary Outcome: Median Duration of Response (DoR) by ICR and Investigator Assessment Using RECIST 1.1
Description: DoR was defined as the time from date of first documented response (which was subsequently confirmed) until date of documented progression or death in the absence of disease progression (i.e. date of progression free survival [PFS] event or censoring - date of first response + 1). The end of response coincided with the date of progression or death from any cause used for the PFS endpoint. The time of initial response was defined as the latest of the dates used towards the first visit that was CR or PR that was subsequently confirmed. If a patient did not progress following a response, the PFS censoring time was used. The Investigator assessment was based on the FAS and the ICR used the EFR analysis set. The median DoR for each assessment is presented and was calculated using the Kaplan-Meier technique.
Time Frame: as for outcome 1
Population: The EFR set included all patients who received at least 1 dose of IP and had measurable disease at baseline according to the independent review of baseline imaging data. The FAS included all patients who received at least 1 dose of either of the IPs.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cediranib + Olaparib
Number analyzed (Participants) | 60
weeks
  ICR assessment (EFR analysis set): number analyzed (Participants) | 59
  ICR assessment (EFR analysis set) | 36.0 [24.4 to 45.0]
  Investigator assessment (FAS) | 45.0 [25.0 to 58.0]

4. Secondary Outcome: Disease Control Rate (DCR) by ICR and Investigator Assessment Using RECIST 1.1
Description: The DCR was defined as the percentage of patients who had a best overall response of CR, PR or Stable Disease (SD) at 6 months.
  CR: Disappearance of all TLs and NTLs since baseline; any pathological lymph nodes selected as TLs must have a reduction in short axis to <10 mm.
  PR: At least a 30% decrease in the sum of the diameters of TL, referencing the baseline sum of diameters.
  SD: Neither sufficient shrinkage of TLs to qualify for PR nor sufficient increase to qualify for progressive disease (PD) (at least a 20% increase in the sum of diameters of TLs with an absolute increase of at least 5 mm and progression of existing NTLs). Patients had to have demonstrated SD for at least 23 weeks following the start of treatment. The Investigator assessment was based on the FAS and the ICR used the EFR analysis set. The percentage of patients with disease control for each assessment is presented.
Time Frame: From baseline up to 6 months after first doses of IPs. RECIST assessments were performed at baseline and every 8 weeks (+/- 1 week) after first doses of IPs until disease progression.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cediranib + Olaparib
Number analyzed (Participants) | 60
percentage of patients
  ICR assessment (EFR analysis set): number analyzed (Participants) | 59
  ICR assessment (EFR analysis set) | 23.7 [13.6 to 36.6]
  Investigator assessment (FAS) | 26.7 [16.1 to 39.7]

5. Secondary Outcome: Median PFS by ICR and Investigator Assessment Using RECIST 1.1
Description: PFS was defined as the time from date of first dose of IP until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdrew from treatment or received another anti-cancer therapy prior to progression (i.e. date of PFS event or censoring - date of first dose + 1). Patients who had not progressed or died at the time of analysis were censored at the time of the latest date of assessment from their last evaluable RECIST assessment.
  The median PFS, calculated using the Kaplan-Meier technique, is presented for the ICR and the Investigator assessment, both based on the FAS.
Time Frame: as for outcome 1
Population: The FAS included all patients who received at least 1 dose of either of the IPs.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cediranib + Olaparib
Number analyzed (Participants) | 60
months
  ICR assessment (FAS) | 5.1 [3.5 to 5.5]
  Investigator assessment (FAS) | 3.8 [3.5 to 6.4]

6. Secondary Outcome: Median Time to Treatment Discontinuation or Death (TDT)
Description: The median time to discontinuation of IPs or death was defined as the time from the date of first dose of IP to the earlier of the date of discontinuation of both IPs, or death date. If 1 IP was discontinued before the other, the TDT reflected the time from the date of first dose to the earliest IP discontinuation date. The median TDT was calculated using the Kaplan-Meier technique.
Time Frame: From baseline to primary analysis DCO (8 months after last patient received their first dose of IPs).
Population: The FAS included all patients who received at least 1 dose of either of the IPs.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cediranib + Olaparib
Number analyzed (Participants) | 60
months | 3.5 [2.7 to 5.1]

7. Secondary Outcome: Median Overall Survival (OS)
Description: OS was defined as the time from the date of first dose of IP until death due to any cause regardless of whether the patient withdrew from treatment or received another anti-cancer therapy (i.e. date of death or censoring - date of first dose + 1). Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive. The median OS was calculated using the Kaplan-Meier technique.
Time Frame: From baseline until death due to any cause, assessed until primary analysis DCO (8 months after last patient received their first dose of IPs).
Population: The FAS included all patients who received at least 1 dose of either of the IPs.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cediranib + Olaparib
Number analyzed (Participants) | 60
months | 13.2 [9.4 to 16.4]

8. Secondary Outcome: Best Observed Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30 Scales
Description: The EORTC QLQ-C30 questionnaire assesses health-related quality of life (HRQoL). The questions are grouped into a global health status/QoL scale, 5 functional scales (physical, role, emotional, cognitive and social), 3 multi-item symptom scales (fatigue, pain, nausea/ vomiting), 5 single items assessing cancer symptoms (dyspnea, loss of appetite, insomnia, constipation, diarrhea), and 1 item on the financial impact of the disease.
  Each scale/item is scored from 0 to 100. Higher scores on the global health status/QoL scale and functional scales indicate better health status/function. Higher scores on the symptom scales/items indicate a greater symptom burden.
  A 10-point change in the score was used to identify patients who improved, stayed the same or deteriorated from baseline. The number of patients with a best observed change from baseline response of improved, stayed the same or deteriorated for each EORTC QLQ-C30 scale/item is presented.
Time Frame: From baseline to primary analysis DCO (8 months after last patient received their first dose of IPs). EORTC QLQ-C30 assessments were performed at baseline and every 8 weeks relative to first dose until discontinuation of IPs.
Population: The FAS included all patients who received at least 1 dose of either of the IPs. Only patients with non-missing baseline and post-baseline data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cediranib + Olaparib
Number analyzed (Participants) | 36
Participants
  Appetite loss: improved | 0
  Appetite loss: stayed the same | 22
  Appetite loss: deteriorated | 14
  Cognitive functioning: improved | 2
  Cognitive functioning: stayed the same | 23
  Cognitive functioning: deteriorated | 11
  Constipation: improved | 2
  Constipation: stayed the same | 27
  Constipation: deteriorated | 7
  Diarrhea: improved | 0
  Diarrhea: stayed the same | 22
  Diarrhea: deteriorated | 14
  Dyspnea: improved | 2
  Dyspnea: stayed the same | 24
  Dyspnea: deteriorated | 10
  Emotional functioning: improved | 2
  Emotional functioning: stayed the same | 31
  Emotional functioning: deteriorated | 3
  Fatigue: improved | 4
  Fatigue: stayed the same | 11
  Fatigue: deteriorated | 21
  Financial difficulties: improved | 2
  Financial difficulties: stayed the same | 32
  Financial difficulties: deteriorated | 2
  Global Health Status / QoL: improved | 1
  Global Health Status / QoL: stayed the same | 19
  Global Health Status / QoL: deteriorated | 16
  Insomnia: improved | 3
  Insomnia: stayed the same | 26
  Insomnia: deteriorated | 7
  Nausea / vomiting: improved | 4
  Nausea / vomiting: stayed the same | 19
  Nausea / vomiting: deteriorated | 13
  Pain: improved | 9
  Pain: stayed the same | 21
  Pain: deteriorated | 6
  Physical functioning: improved | 0
  Physical functioning: stayed the same | 24
  Physical functioning: deteriorated | 12
  Role functioning: improved | 1
  Role functioning: stayed the same | 18
  Role functioning: deteriorated | 17
  Social functioning: improved | 1
  Social functioning: stayed the same | 22
  Social functioning: deteriorated | 13

9. Secondary Outcome: Best Observed Change From Baseline in EORTC QLQ-OV28
Description: The EORTC QLQ-OV28 is specific for ovarian cancer and consists of 28 items assessing abdominal/gastrointestinal symptoms (6 items), peripheral neuropathy (2 items), other chemotherapy side effects (5 items), hormonal symptoms (2 items), body image (2 items), attitudes to disease/treatment (3 items), sexuality (4 items) and 4 other single items.
  Each scale was scored from 0 to 100 with higher scores on the symptom scales indicating greater symptom burden.
  The best observed change from baseline is presented for each EORTC QLQ-OV28 scale, where a 10-point change in the score was used to identify patients who improved, stayed the same or deteriorated. The number of patients with a best observed change from baseline response of improved, stayed the same, or deteriorated in the EORTC QLQ-OV28 is presented.
Time Frame: From baseline to primary analysis DCO (8 months after last patient received their first dose of IPs). EORTC QLQ-OV28 assessments were performed at baseline and every 8 weeks relative to first dose until discontinuation of IPs.
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cediranib + Olaparib
Number analyzed (Participants) | 32
Participants
  Abdominal / Gastrointestinal: improved | 2
  Abdominal / Gastrointestinal: stayed the same | 18
  Abdominal / Gastrointestinal: deteriorated | 12
  Attitude to disease / treatment: improved | 3
  Attitude to disease / treatment: stayed the same | 16
  Attitude to disease / treatment: deteriorated | 13
  Body image: improved | 7
  Body image: stayed the same | 19
  Body image: deteriorated | 6
  Chemotherapy side effects: improved | 1
  Chemotherapy side effects: stayed the same | 24
  Chemotherapy side effects: deteriorated | 7
  Hormonal: improved | 2
  Hormonal: stayed the same | 25
  Hormonal: deteriorated | 5
  Other single items: improved | 1
  Other single items: stayed the same | 19
  Other single items: deteriorated | 12
  Peripheral neuropathy: improved | 1
  Peripheral neuropathy: stayed the same | 24
  Peripheral neuropathy: deteriorated | 7
  Sexuality: improved | 2
  Sexuality: stayed the same | 26
  Sexuality: deteriorated | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected with an onset date on or after the date of first dose of IP and up to and including 30 days following the date of last dose of IP. Assessed until primary analysis DCO (over a period of approximately 2 years and 7 months).
Description: The safety analysis set included all patients who received at least 1 dose of either IP.
Arm/Group | Cediranib + Olaparib
All-Cause Mortality (participants affected / at risk) | 36/60
Serious Adverse Events (participants affected / at risk) | 22/60
Other Adverse Events (participants affected / at risk) | 56/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cediranib + Olaparib (N=60)
Anaemia (Blood and lymphatic system disorders) | 1 (2)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Oedema peripheral (General disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1)
Hepatic encephalopathy (Hepatobiliary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cediranib + Olaparib (N=60)
Anaemia (Blood and lymphatic system disorders) | 12 (19)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (15)
Hypothyroidism (Endocrine disorders) | 9 (9)
Abdominal distension (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 20 (27)
Constipation (Gastrointestinal disorders) | 17 (19)
Diarrhoea (Gastrointestinal disorders) | 40 (78)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 39 (50)
Oral pain (Gastrointestinal disorders) | 6 (6)
Stomatitis (Gastrointestinal disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 23 (38)
Asthenia (General disorders) | 6 (9)
Fatigue (General disorders) | 41 (50)
Mucosal inflammation (General disorders) | 5 (8)
Oedema peripheral (General disorders) | 9 (11)
Urinary tract infection (Infections and infestations) | 10 (11)
Aspartate aminotransferase increased (Investigations) | 6 (7)
Blood alkaline phosphatase increased (Investigations) | 5 (6)
Blood creatinine increased (Investigations) | 9 (11)
Blood thyroid stimulating hormone increased (Investigations) | 7 (7)
Platelet count decreased (Investigations) | 7 (8)
Weight decreased (Investigations) | 8 (9)
Decreased appetite (Metabolism and nutrition disorders) | 21 (24)
Dehydration (Metabolism and nutrition disorders) | 10 (15)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 15 (25)
Hyponatraemia (Metabolism and nutrition disorders) | 12 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (8)
Dizziness (Nervous system disorders) | 7 (8)
Dysgeusia (Nervous system disorders) | 11 (12)
Headache (Nervous system disorders) | 21 (26)
Neuropathy peripheral (Nervous system disorders) | 7 (7)
Anxiety (Psychiatric disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 5 (6)
Proteinuria (Renal and urinary disorders) | 7 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (13)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (22)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Hypertension (Vascular disorders) | 39 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and the PI are entitled to publish the results of or make presentations related to the study, provided that any publication or presentation to be made within 2 years of study completion require the Company's prior written consent. All publications or presentations shall be consistent with academic standards and International Committee of Medical Journal Editors guidelines, not be false or misleading, comply with all Applicable Laws and not be made for any commercial purpose.

DOCUMENTS (2):
  • Study Protocol (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT02889900/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT02889900/SAP_001.pdf